CLINICAL TRIAL: NCT00423540
Title: Magnesium Status & Effect of Magnesium Infusions on Rest Cramps
Brief Title: Exploring the Role of Magnesium in Rest Cramps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Dr. Scott Garrison, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H06-03345; Health Canada #9427-R1243-21C
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2008-12-10 (Estimated); Status verified 2008-12

CONDITIONS: Rest Cramps
Keywords: magnesium infusion; magnesium sulfate; rest cramps; nocturnal leg cramps; muscle cramps; fractional urinary excretion; urinary excretion; 24 hour urine; serum magnesium; magnesium deficiency; family practice; general practice; richmond; cramp frequency; magnesium status; urinary magnesium; cramp diary; sf 36
MeSH Terms: conditions — Sleep-Wake Transition Disorders; Muscle Cramp; Magnesium Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Intravenous Infusion of Magnesium Sulfate — See Detailed Description.

SUMMARY:
This study sets out to show whether infusions of magnesium can lessen the frequency of rest cramps and to determine whether rest cramp sufferers have a deficiency in magnesium.

DETAILED DESCRIPTION:
Subjects will be randomized to receive 5 days of 4 hour IV infusions of D5W either with or without 20 mmol magnesium sulfate added. Twenty four hour urinary excretion of magnesium will be determined on the first day of infusions to assess whether magnesium deficiency is present. Ten normal controls will also undergo a single infusion and collection of urine to serve as a comparison group for the urinary excretion data.

ELIGIBILITY:
Inclusion Criteria:

* ≥2 leg or foot cramps per week in a 4 week run-in diary

Exclusion Criteria:

* eGFR<50
* Neurologic disease
* Pregnancy
* Heart block
* Bradyarhythmia without pacemaker
* Digoxin use
* Liver disease
* Addison's disease
* History of MI
* CHF
* Absence of detectable reflexes

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of leg cramps per week (active versus placebo) over the first 30 days post infusions compared to the 30 days prior to randomization (as recorded in patient diaries). | See above

SECONDARY OUTCOMES:
Assessment of magnesium status at trial entry as determined by 24 hour fractional excretion of magnesium on day 1 of infusions.
Subjective assessment as to whether cramps were unchanged, more, or less frequent /painful/"bothersome" over the 3 months. following infusions. | See above
Overall quality of life changes as measured by an SF36 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Garrison Scott, MD, Principal Investigator — University of British Columbia
Locations (1):
- Richmond Hospital, Richmond, British Columbia, Canada